CLINICAL TRIAL: NCT00651820
Title: A Randomized, Double-blind, Paired-Comparison of the Effect of Collagenase Santyl® Ointment on Healing and Scarring Characteristics of 600μm Dermatome Wounds
Brief Title: Effect of Collagenase on Healing and Scarring
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Healthpoint (Industry)
Responsible Party: Shai M. Rozen, MD, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 017 101 09 001
Record Dates: First submitted 2008-03-20; First posted 2008-04-03 (Estimated); Results first posted 2011-01-26 (Estimated); Last update posted 2011-06-09 (Estimated); Status verified 2011-06

CONDITIONS: Scarring; Impaired Wound Healing
Keywords: wound healing; scarring; collagenase; Santyl
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Collagenase Santyl Rate of Wound Closure (Experimental): Dermatome-induced skin wounds treated with drug active (collagenase).
  Interventions: Drug: Collagenase Santyl
- Vehicle Rate of Wound Closure (Placebo Comparator): Dermatome-induced skin wounds treated with Vehicle alone.
  Interventions: Drug: Collagenase Santyl Vehicle

INTERVENTIONS:
Drug: Collagenase Santyl — Dermatome-induced skin wounds treated with drug active.
  Each subject serves as his own control receiving both treatments in parallel.
  Arms: Collagenase Santyl Rate of Wound Closure
Drug: Collagenase Santyl Vehicle — Dermatome-induced skin wounds treated with Vehicle alone. Each subject serves as his own control receiving both treatments in parallel.
  Arms: Vehicle Rate of Wound Closure

SUMMARY:
A study to compare the rate of complete wound closure and quality of resulting scar at 3, 6 and 9 months, between dermatome-induced skin wounds treated with Collagenase Santyl Ointment versus vehicle alone.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent
2. Willing to attend all required study visits

Exclusion Criteria:

1. Known hypersensitivity to Clostridial collagenase
2. Anticoagulants (blood thinners, including aspirin) within two weeks
3. Congenital skin disorder which affects keratinocytes, elastin, or collagen
4. Any dermatologic disease which may be aggravated or provoked by the wounding procedure
5. Dark skin pigmentation to a degree which is very likely to obscure the assessment of vascularization post-wounding
6. At risk of keloid or hypertrophic scar formation
7. Scars, tattoos or deformities (i.e., contractures) on the inner aspect of the upper arm area where the wound will be placed
8. Any skin disorder which causes delayed healing
9. Disrupted lymphatic drainage of the arm to be studied, or previously diagnosed thoracic outlet syndrome
10. Taking concomitant medications at doses which are known to interfere with healing, such as non-steroidal anti-inflammatory drugs, anti-neoplastic drugs, or immunosuppressive drugs

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2008-04; Primary Completion 2009-11 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herbert B Slade, MD, Study Director — Healthpoint
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Rate of Wound Closure Collagenase Santyl vs. Vehicle: Dermatome-induced skin wounds treated with drug active (collagenase). Each subject received 2 identical wounds, one on each arm. One arm was treated with Collagenase Santyl, the other with Vehicle. Each subject acted as their own control.
Period: Overall Study
Arm/Group | Rate of Wound Closure Collagenase Santyl vs. Vehicle
Started | 28
Completed | 26
Not Completed | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Arm/Group | Rate of Wound Closure Collagenase Santyl vs. Vehicle
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 28
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 37.6 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Time to Complete Wound Closure Collagenase Santyl and Vehicle
Time Frame: 21 days
Population: Analysis was performed on all subjects as intent-to-treat (ITT).
Measure: Mean (95% Confidence Interval); unit: Days
Units Other Than Participants: Dermatome-induced wounds on Arms
Groups:
- Collagenase Santyl Rate of Wound Closure: Dermatome-induced skin wounds treated with drug active (collagenase). Each subject received 2 identical wounds, one on each arm. One arm was treated with Collagenase Santyl, the other with Vehicle. Each subject acted as their own control.
- Vehicle Rate to Complete Wound Healing: Dermatome-induced skin wounds treated with Vehicle alone. Each subject received 2 identical wounds, one on each arm. One arm was treated with Collagenase Santyl, the other with Vehicle. Each subject acted as their own control.
Arm/Group | Collagenase Santyl Rate of Wound Closure | Vehicle Rate to Complete Wound Healing
Number analyzed (Participants) | 28 | 28
Number analyzed (Dermatome-induced wounds on Arms) | 28 | 28
Days | 12.9 [6 to 26] | 13.0 [8 to 26]
Statistical Analysis 1: Comparison: Collagenase Santyl Rate of Wound Closure vs Vehicle Rate to Complete Wound Healing; Each subject served as their own control, each receiving duplicate dermatome-induced wounds with 1 wound treated with active drug and the other treated with vehicle. Mean time to wound closure was calculated for the wounds treated with drug, the wounds treated with vehicle, and an over-all mean time to wound closure; Test type: Superiority or Other; p < 0.05, Paired-Prentice Wilcoxon (PPW); Time to complete wound closure Drug(T1)and Vehicle(T2)Hypothesis, Ho: T1=T2,using paired Prentice-Wilcoxon at significant level of 5%, 2-sided

2. Secondary Outcome: Differences in Scar Viscoelasticity Between Wounds Treated With Collagenase Santyl and Its Vehicle
Description: Differences in Scar Viscoelasticity between wounds treated with Collagenase Santyl and its vehicle as measured by Stiffness and Energy Absorption using BTC-2000 measurements.
Time Frame: 9 Months
Population: Analysis performed on Intent-to-Treat (ITT) population
Measure: Mean (Standard Deviation); unit: mmHg/mm
Units Other Than Participants: Dermatome-induced wounds on Arms
Groups:
- Vehicle Rate of Wound Closure: Dermatome-induced skin wounds treated with Vehicle alone. Each subject received 2 identical wounds, one on each arm. One arm was treated with Collagenase Santyl, the other with Vehicle. Each subject acted as their own control.
Arm/Group | Collagenase Santyl Rate of Wound Closure | Vehicle Rate of Wound Closure
Number analyzed (Participants) | 28 | 28
Number analyzed (Dermatome-induced wounds on Arms) | 28 | 28
mmHg/mm
  Stiffness | 184.25 (37.47) | 174.05 (46.51)
  Energy Absorption | 72.6 (18.33) | 78.48 (24.96)
Statistical Analysis 1: Comparison: Collagenase Santyl Rate of Wound Closure vs Vehicle Rate of Wound Closure; Stiffness: Paired t-test and Wilcoxon signed rank test were used for testing any significant differences (Sig. diff.) between the two treatments; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = 10.20
Statistical Analysis 2: Comparison: Collagenase Santyl Rate of Wound Closure vs Vehicle Rate of Wound Closure; Energy Absorption: Paired t-test and Wilcoxon signed rank test were used for testing any significant differences (Sig. diff.) between the two treatments; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Final Values) = -5.88

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the 9 month period of the study
Description: Adverse events were captured, but the Investigator did not always capture which arm exhibited the adverse event, so no in depth analysis could be performed. Of the 2 subjects whose adverse event was probably related to test article (as designated by the Investigator), only 1 had the arm designated and that arm was treated with vehicle.
Arm/Group | Rate of Wound Closure Collagenase Santyl vs. Vehicle
Serious Adverse Events (participants affected / at risk) | 1/28
Other Adverse Events (participants affected / at risk) | 4/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rate of Wound Closure Collagenase Santyl vs. Vehicle (N=28)
Brain Aneurysm (Vascular disorders) | 1 (1) — The 1 SAE (brain aneurysm) was reported as severe and was unrelated to the test articles
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rate of Wound Closure Collagenase Santyl vs. Vehicle (N=28)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) — Wound redness (erythema)- Investigator specified Right Arm for 1 subject, which was treated with Vehicle. Investigator did not specify arm for the second subject with erythema, so causative agent could not be determined.
Rash (Skin and subcutaneous tissue disorders) | 2 (2) — For 1 subject the Investigator did not specify which arm developed the rash, so unable to determine if Collagenase Santyl or its vehicle was causative agent. For the other subject the Investigator specified that both arms developed a rash.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No